CLINICAL TRIAL: NCT05804734
Title: Vitamin K Antagonist Versus Direct Oral Anticoagulant Treatments in Hemophilia
Acronym: KADOAH
Status: Completed | Type: Observational
Sponsor: Groupe Maladies hémorragiques de Bretagne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_VKA-DOA_01
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Hemophilia A; Hemophilia B; Anticoagulant-induced Bleeding
Keywords: Hemophilia A; Hemophilia B; Anticoagulant-induced Bleeding
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Cases: Patients with hemophilia receiving an anticoagulant treatment in the period 2012-2021
  Interventions: Drug: Vitamin K Antagonist - Drug
- Controls: Patients with hemophilia cross-matched with cases on the age, the hemophilia's severity, the hemophilia's type, and the HAS-BLED score.

INTERVENTIONS:
Drug: Vitamin K Antagonist - Drug — Only clinical data (number and types of severe bleeding events, HAS-BLED score, CHA2DS2-VASc score) are collected during the follow-up:
  * For cases when they received an anticoagulant treatment and during the 12 months preceding this treatment,
  * For controls during the same periods of their cross-matched cases when reciving anticoagulant treatment.
  Other Names: direct oral anticoagulant
  Groups: Cases

SUMMARY:
Hemophilia is a rare X-linked bleeding disorder responsible for deficiency of coagulation factor VIII (FVIII) or IX (FIX). The main clinical manifestation is increased bleeding throughout the life which is directly correlated to the severity of the hemophilia, either mild (FVIII/FIX: 6-40), moderate (FVIII/FIX: 1-5%), or severe (FVIII/FIX<1%). Thanks to new therapies and long-term specialized follow-up by hemophilia treatment centers (HTCs), the life expectancy of patients with hemophilia (PWH) has improved considerably, even reaching that of the general population (1).

Healthcare professionals are so more confronted to PWH with age-related pathologies, in particular cardiovascular pathologies such as atrial fibrillation, acute coronary syndromes or thromboembolic events (arterial or venous). It is now recommended in PWH that an anticoagulant treatment (AC) be prescribed as in the general population (2,3,4). The recently published COCHE study demonstrated a significantly increased risk of bleeding in PWH receiving antithrombotic treatment. This bleeding risk depended significantly on the type of antithrombotic treatment, which was higher for anticoagulant vs antiplatelet drugs, on basal levels of FVIII or FIX, and on the HAS-BLED score (5).

Nowadays in the general population, among anticoagulant drugs, direct oral anticoagulants (DOACs) are preferred to vitamin K antagonist (KVA), thanks to their reduced risk of bleeding particularly intracerebral bleeding and better anticoagulant stability over time (6). However, we do not yet know precisely whether DOACs could occupy the same place in the PWH population because of the lack of evidence-based data due to the very small number of these patients, although some authors already recommend them over KVA. The KADOAH study was therefore set up to try to provide initial elements for future recommendations. Its main objective was to compare the level of bleeding risk of PWH treated with VKA vs DOACs.

DETAILED DESCRIPTION:
The KADOAH study is an observational, retrospective and multicenter case-control study conducted in Hemophilia Treatment Centers (HTC) of the French Grand-Ouest interregion including HTCs of Brest, Caen, Le Mans, Nantes, Rennes and Rouen.

Objectives of the KADOAH study are:

* To compare the risk of bleeding events of 2 types of long-term anticoagulant treatment, vitamin K antagonists (VKA) versus Direct Oral Anticoagulants (DOAC), in patients with hemophilia,
* To describe the different types of bleeding events that occur during anticoagulant treatments in patients with hemophilia,
* To investigate for the influence of the HAS-BLED score on the risk of bleeding events in patients with hemophilia receiving a long-term anticoagulant treatment.

Inclusion criteria:

* Cases :
* Males at any ages with hemophilia of any severity and of any type,
* Patients having received or receiving a long-term anticoagulant treatment (during at least 6 consecutive months) during the period from 2012 to 2021,
* Regular follow-up in a hemophilia treatment center.
* Controls cross-matched with cases on :
* Age (+/- 5 years),
* Hemophilia type (either A or B)
* Hemophilia severity (for mild hemophilia: same basal factor level +/- 5%),
* HAS-BLED score (same score +/- 1).

Exclusion criteria:

* Lost to medical follow-up,
* Refusal to participate in the study,
* Unable to understand the study's French letter of non-opposition and information.

Collected data:

All data collected in this study were issued from the medical files at the moment of the inclusion in the study. They include:

* The age,
* The hemophilia's type,
* The hemophilia's severity and last basal factor VIII or IX level,
* The treatment with anticoagulant drug for cases including :
* Type of drug (either VKA or DOAC)
* Duration of treatments
* Treatments dosages,
* Compliance of treatments,
* Indications,
* If stopped prematurely, reasons for stopping.
* The occurrence of severe bleeding events (SBE) following the ISTH definition (7):
* The number of SBE per patient,
* The types of SBE,
* The treatment of SBE.
* The HAS-BLED score calculated with the presence or absence of the following items:
* High arterial pressure,
* Abnormal renal and/or liver functions,
* Hemorrhagic stroke,
* Bleeding antecedent,
* Age >65 years,
* Treatments altering the hemostasis (out of the anticoagulants) and/or alcohol intoxication.
* The CHA2DS-VASc score calculated with the presence or absence of the following items:
* Cardiac insufficiency/left ventricular dysfunction,
* High arterial pressure,
* Age ≥ 75 years, or age = 65 - 74 years,
* Diabetes,
* History of thrombotic events (transient ischemic cerebral attack or stroke, venous thromboembolic events)
* Associated treatment with a proton pomp inhibitor or other gastric protector,

Statistical analyses Descriptive characteristics were analyzed with median values, their 25-75% interquartile ranges (IQR) and minimum-maximum values (MIN-MAX), or mean values with standard deviation (SD). The Fisher's exact test will be performed to compare proportions in contingency tables and the t Student test to compare continuous variables. An approximate 95% confidence interval will be determined (95% CI) for every statistical analysis and a p-value <0.05 will be considered statistically significant. The GraphPad v7.0 (Prism Software Inc. San Diego CA) will be used to perform the statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Cases :

  * Males at any ages with hemophilia of any severity and of any type,
  * Patients having received or receiving a long-term anticoagulant treatment (during at least 6 consecutive months) during the period from 2012 to 2021,
  * Regular follow-up in a hemophilia treatment center.
* Controls : patients with hemophilia cross-matched with cases on:

  * Age (+/- 5 years),
  * Hemophilia type (either A or B)
  * Hemophilia severity (for mild hemophilia: same basal factor level +/- 5%),
  * HAS-BLED score (same score +/- 1).

Exclusion Criteria:

* Lost to medical follow-up,
* Refusal to participate in the study,
* Unable to understand the study's French letter of non-opposition and information.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes only patients with hemophilia: cases who are patients having received an anticoagulant treatment (cases) for at least 6 months during the period 2112-2021, and controls without anticoagulant treatment cross-matched with cases on the age, the severity and type of hemophilia, and the HAS-BLED score.
  All the data collected in this study are issued from the medical files.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the number of severe bleeding events occurring in patients with hemophilia receiving a vitamin K antagonist treatment versus patients with hemophilia receiving a direct oral anticoagulant treatment. | All over the duration of the anticoagulant treatment in the period 2012-2021
  Number of severe bleeding events

SECONDARY OUTCOMES:
Comparison of the number of severe bleeding events occurring in patients with hemophilia receiving an anticoagulant treatment versus their cross-matched controls not receiving an anticoagulant treatment. | All over the duration of the anticoagulant treatment in the period 2012-2021
  Number of severe bleeding events
Description of the types of severe bleeding events occurring in patients with hemophilia receiving an anticoagulant treatment (either vitamin K antagonist or direct oral anticoagulant treatment). | All over the duration of the anticoagulant treatment in the period 2012-2021
  Types of bleeding
The influence of the HAS-BLED score on the risk of severe bleeding events in patients with hemophilia receiving an anticoagulant treatment. | All over the duration of the anticoagulant treatment in the period 2012-2021
  HAS-BLED score
The influence of a treatment with proton pomp inhibitor on the risk of gastrointerstinal bleeding events in patients with hemophilia receiving an anticoagulant treatment. | All over the duration of the anticoagulant treatment in the period 2012-2021
  Number of gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Benoît GUILLET, MD PhD, Study Director — University hospital of rennes, France
Locations (6):
- France (6):
  - Hemophilia treatment center of Brest, Brest
  - Hemophilia treatment center of caen, Caen
  - Hemophilia treatment center of Le Mans, Le Mans
  - Hemophilia treatment center of Nantes, Nantes
  - Hemophilia treatment center of Rennes, Rennes
  - Hemophilia treatment center of Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade JG, Verma A, Mitchell LB, Parkash R, Leblanc K, Atzema C, Healey JS, Bell A, Cairns J, Connolly S, Cox J, Dorian P, Gladstone D, McMurtry MS, Nair GM, Pilote L, Sarrazin JF, Sharma M, Skanes A, Talajic M, Tsang T, Verma S, Wyse DG, Nattel S, Macle L; CCS Atrial Fibrillation Guidelines Committee. 2018 Focused Update of the Canadian Cardiovascular Society Guidelines for the Management of Atrial Fibrillation. Can J Cardiol. 2018 Nov;34(11):1371-1392. doi: 10.1016/j.cjca.2018.08.026. PMID 30404743
- [Background] Ferraris VA, Boral LI, Cohen AJ, Smyth SS, White GC 2nd. Consensus review of the treatment of cardiovascular disease in people with hemophilia A and B. Cardiol Rev. 2015 Mar-Apr;23(2):53-68. doi: 10.1097/CRD.0000000000000045. PMID 25436468
- [Background] Schutgens RE, van der Heijden JF, Mauser-Bunschoten EP, Mannucci PM. New concepts for anticoagulant therapy in persons with hemophilia. Blood. 2016 Nov 17;128(20):2471-2474. doi: 10.1182/blood-2016-07-727032. Epub 2016 Sep 26. No abstract available. PMID 27670425
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Result] Darby SC, Kan SW, Spooner RJ, Giangrande PL, Hill FG, Hay CR, Lee CA, Ludlam CA, Williams M. Mortality rates, life expectancy, and causes of death in people with hemophilia A or B in the United Kingdom who were not infected with HIV. Blood. 2007 Aug 1;110(3):815-25. doi: 10.1182/blood-2006-10-050435. Epub 2007 Apr 19. PMID 17446349
- [Result] Guillet B, Cayla G, Lebreton A, Trillot N, Wibaut B, Falaise C, Castet S, Gautier P, Claeyssens S, Schved JF. Long-Term Antithrombotic Treatments Prescribed for Cardiovascular Diseases in Patients with Hemophilia: Results from the French Registry. Thromb Haemost. 2021 Mar;121(3):287-296. doi: 10.1055/s-0040-1718410. Epub 2020 Oct 24. PMID 33099283
- [Result] Gomez-Outes A, Terleira-Fernandez AI, Calvo-Rojas G, Suarez-Gea ML, Vargas-Castrillon E. Dabigatran, Rivaroxaban, or Apixaban versus Warfarin in Patients with Nonvalvular Atrial Fibrillation: A Systematic Review and Meta-Analysis of Subgroups. Thrombosis. 2013;2013:640723. doi: 10.1155/2013/640723. Epub 2013 Dec 22. PMID 24455237